CLINICAL TRIAL: NCT01721460
Title: Effects of Dexmedetomidine on Neuronal Activity in the Subthalamic Nucleus During Deep Brain Stimulation (DBS) Electrode Implantation Surgery
Brief Title: Effects of Dexmedetomidine on Activity in the Subthalamic Nucleus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0400
Record Dates: First submitted 2012-10-30; First posted 2012-11-05 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Parkinson's Disease; Deep Brain Stimulation Surgery
Keywords: SubThalamic Nucleus; Microelectrode recording; Deep Brain Stimulation Electrode implantation
MeSH Terms: conditions — Parkinson Disease | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexmedetomidine during MER (Experimental): The study is performed in patients undergoing DBS electrode implantation to their STN for the treatment of parkinson's disease. Microelectrode recording (MER) is performed as part of STN electrode implantation surgery, to increase the precision of the stimulating electrode placement. The study includes administration of dexmedetomidine while recording electrical activity at a single location to evaluate the effects of this drug on the MER.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine infusion will be started with a loading dose of 1 mcg/Kg over ten to 20 minutes followed by a maintenance infusion of 0.7 mcg/Kg/hr until stable sedation is achieved.
  Other Names: Precedex

SUMMARY:
The purpose of this research study is to find out whether dexmedetomidine changes brain cell activity in the subthalamic nucleus (STN).

DETAILED DESCRIPTION:
In order to find whether dexmedetomidine is optimal for sedation during Deep brain stimulation surgery, we will measure the electrical activity in the STN during Deep brain stimulation surgery, and measure how this activity is changed during administration of Dexmedetomidine. We hypothesize that dexmedetomidine does not change the firing rate and pattern in the STN.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo bilateral STN electrode implantation surgery with Micro-electrode recording for the treatment of Parkinson's disease.

Exclusion Criteria:

* Hypersensitivity to dexmedetomidine
* Bradycardia: Sinus rhythm slower than 50 bpm
* Known or suspected obstructive sleep apnea
* Suspected difficult intubation
* Pregnancy
* Under 18 years of age or over 85 years of age
* Cognitive disability impairing understanding the experiment or signing the informed consent form

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aeyal Raz, MD, PhD, Principal Investigator — University of Wisconsin, Madison, Department of anesthesiology
Locations (1):
- University of Wisconsin - Madison, School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amlong C, Rusy D, Sanders RD, Lake W, Raz A. Dexmedetomidine depresses neuronal activity in the subthalamic nucleus during deep brain stimulation electrode implantation surgery. BJA Open. 2022 Sep 9;3:100088. doi: 10.1016/j.bjao.2022.100088. eCollection 2022 Sep. PMID 37588575

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine During MER: Administration of dexmedetomidine during the Microelectrode recording (MER) part of subthalamic nucleus (STN) electrode implantation surgery.
  Dexmedetomidine: Dexmedetomidine infusion will be started with a loading dose of 1 mcg/Kg over ten to 20 minutes followed by a maintenance infusion of 0.7 mcg/Kg/hr until stable sedation is achieved.
Period: Overall Study
Arm/Group | Dexmedetomidine During MER
Started | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Dexmedetomidine During MER: Administration of dexmedetomidine during the Microelectrode recording part of STN electrode implantation surgery.
  Dexmedetomidine: Dexmedetomidine infusion will be started with a loading dose of 1 mcg/Kg over ten to 20 minutes followed by a maintenance infusion of 0.7 mcg/Kg/hr until stable sedation is achieved.
Arm/Group | Dexmedetomidine During MER
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 61.5 [53 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Population Spiking Activity
Description: We calculated the root mean square (RMS) of the high frequency electrical activity. This is a common measure for the spiking rate of the population of neurons in the vicinity of the electrode tip. This Measure has been previously described as a useful measure to determine the target location during deep brain stimulation (DBS) procedures. We calculated the change in RMS inside the STN between baseline and peak sedation.
  For each subject we normalized the RMS to the RMS of the electrical activity outside the nucleus. This is done to eliminate the effects of noise and variability in electrode resistance. Thus, the normalized RMS is a pure number with no units.
Time Frame: 20-35 minutes following drug administration
Population: All participants had the normalized RMS of the electrical activity calculated during control period, and under maximal sedation, and the difference between the two was calculated and normalized.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Dexmedetomidine Modulation of MER: Change in RMS value between baseline (awake) and maximal sedation during dexmedetomidine administration.
Arm/Group | Dexmedetomidine Modulation of MER
Number analyzed (Participants) | 5
Percent change | 42.8 (12.7)

2. Secondary Outcome: Change in Average Firing Pattern in the STN
Description: We've used total power in the Beta range (13-30Hz) to evaluate change in firing pattern and oscillation frequency.
Time Frame: 20-35 minutes following drug administration
Population: All participants that received sedation
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Dexmedetomidine During MER
Number analyzed (Participants) | 5
percentage change | 39.9 (76.2)

3. Secondary Outcome: Time to Recovery
Description: The time it takes for the patient to become alert after drug administration is stopped.
Time Frame: 20-60 minutes after stopping drug administration
Population: All participants that received sedation.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Dexmedetomidine During MER: Administration of dexmedetomidine during the Microelectrode recording (MER) part of subthalamic nucleus (STN) electrode implantation surgery.
Arm/Group | Dexmedetomidine During MER
Number analyzed (Participants) | 5
minutes | 16 (13)

4. Secondary Outcome: Portion of Participants With Timely Return of the Neuronal Activity to Baseline
Description: The portion of patients in which neuronal activity returned to baseline within 30 after stopping sedation.
Time Frame: 30 minutes after stopping drug administration
Population: All participants that received sedation. As the activity did not return to baseline within the allocated time for the study (30 minutes), we report the portion of patients in which the activity returned to baseline within this time.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexmedetomidine During MER
Number analyzed (Participants) | 5
Participants | 2

ADVERSE EVENTS:
Time Frame: Duration of procedure, 6-10 hours.
Groups:
- Treatment: Administration of dexmedetomidine during the Microelectrode recording part of STN electrode implantation surgery.
  Dexmedetomidine: Dexmedetomidine infusion will be started with a loading dose of 1 mcg/Kg over ten to 20 minutes followed by a maintenance infusion of 0.7 mcg/Kg/hr until stable sedation is achieved.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes